CLINICAL TRIAL: NCT03863678
Title: Effects of Dry Needling on Spasticity, Upper and Lower Extremity Functions, Balance and Independence Level in Addition to Neurodevelopmental Therapy in Patients With Stroke
Brief Title: Effects of Dry Needling on Spasticity, Functions, Balance and Independence Level in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Kübra Küçüktepe, Msc Physiotherapist, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KK 1695
Record Dates: First submitted 2019-02-24; First posted 2019-03-05 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Stroke; CVA (Cerebrovascular Accident)
Keywords: dry needling; neurodevelopmental therapy; spasticity; balance; functions; independence
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodevelopmental therapy (Experimental): Group 1 will only receive Neurodevelopmental therapy (NDT), for 12 sessions.
  Interventions: Other: Neurodevelopemental therapy (NDT)
- Neurodevelopemental therapy and dry needling therapy (Experimental): Group 2 will receive Neurodevelopmental therapy (NDT) and dry needling therapy, for 12 sessions.
  Interventions: Other: Neurodevelopemental therapy (NDT) and dry needling

INTERVENTIONS:
Other: Neurodevelopemental therapy (NDT) — NDT treatment will be given for 45 minutes, 3 sessions per week in 4 weeks period (total of 12 sessions).
  Arms: Neurodevelopmental therapy
Other: Neurodevelopemental therapy (NDT) and dry needling — NDT treatment will be given for 45 minutes, 3 sessions per week in 4 weeks period (total of 12 sessions). Dry needling will be applied on M. Gastrocnemius, M.Quadriceps, M.Flexor Carpi Radialis, and M.Biceps Brachii muscles, 60 seconds (sec) for each muscle groups at the end of the NDT treatment.
  Arms: Neurodevelopemental therapy and dry needling therapy

SUMMARY:
The aim of this study is to investigate the effects of dry needling method in addition to neurodevelopmental therapy on spasticity, upper and lower extremity functions, balance and independence level in patients with stroke who have spasticity.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of dry needling method in addition to neurodevelopmental therapy on spasticity, upper and lower extremity functions, balance and independence level in patients with stroke who have spasticity. In this study, goniometric measurement, Modified Ashworth Scale, Nine Hole Peg Test, 10 Meter Walking Test, Fullerton Advanced Balance Scale and Functional Independence Scale will be used for outcome measurement. The participants will be randomised into two groups; Group 1 will receive NDT and Group 2 will receive both NDT and dry needling therapy. Both groups will be given 45 minutes of NDT, 3 sessions per week in 4 weeks period (total of 12 sessions). Group 2 will also receive dry needling therapy 3 sessions per week in 4 weeks period (total of 12 sessions). Dry needling will be applied on M. Gastrocnemius, M.Quadriceps, M.Flexor Carpi Radialis and M.Biceps Brachii muscles. The application time on each muscle will be 60 seconds (sec). Fast in and fast out technique will be used for dry needling therapy. All patients will be measured before treatment (T1) and after treatment (T3). An inter-measurement will be performed after the treatment session (T2) in addition to T1 and T3 measurements in the Group 2, to evaluate the acute effects of dry needling therapy. No additional treatment will be applied to the Group 1. All assessments will be performed by the same physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* First time stroke,
* Patients who has spasticity due to stroke,
* At least 6 months after stroke,
* Individuals between the ages of 18-75 will be included in the study.

Exclusion Criteria:

* Any contraindication for dry needling (eg, anticoagulants, infections, bleeding, etc.),
* Having diabetes,
* Having cardiovascular diseases,
* Having any other neurological problems,
* Application of Botox within 6 months prior to the study,
* Individuals included in another treatment program will not be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-05-12 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Range of movement (ROM) measurement | Change from baseline ROM measurement at 4 weeks
  Measurement of joint movement of individuals will be done by a goniometer by the same physiotherapist. First passive normal joint movement then active normal joint movement will be evaluated and recorded.
Modified Ashworth Scale (MAS) | At the baseline and at the end of 4 weeks
  Modified ashworth scale (MAS) will be used to evaluate the spasticity of upper (elbow flexors flexor carpi radialis) and lower (quadriceps and gastrocnemius) extremity muscles. The MAS assess the level of spasticity on ordinal scale from 0 to 4 based on the level of resistance in response to a quick and passive movement. According to the MAS scale, 0 represents no increase in muscle tone, 1 represents slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension, 1+ represents increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM, 2 represents more marked increase in muscle tone through most of the ROM, but affected part(s) easily moved, 3 represents considerable increase in muscle tone, passive movement difficult and 4 represents affected part(s) rigid in flexion or extension.

SECONDARY OUTCOMES:
Nine Hole Peg Test | At the baseline and at the end of 4 weeks
  NHPT (Nine Hole Peg Test); It is a time test in which the thin hand skill is quantitatively measured. During the test, the patient sits on the table where the nine hole board is located and closes the empty hole with the wooden or plastic bars.
10 Meter Walking Test | At the baseline and at the end of 4 weeks
  The walking speed of the patients will be measured with a ten-meter walking test (10MWT). The walking time of the patient in 10 meters is recorded in seconds and the walking speed in m / s is calculated.
Fullerton Advanced Balance Scale | At the baseline and at the end of 4 weeks
  He will use a total of 10 items of balance scale to assess the balance of the patients. Each item is rated between 0-4. It will be evaluated over 40 points.
Functional Independence Scale | At the baseline and at the end of 4 weeks
  It is a generic and global activity scale and shows how independent it is in daily basic, physical and cognitive activities.Each item is scored at seven levels (1-7), Level 1: Total Assistance, Level 7: Indicates full independence. The total FIM score may vary between 18-126. FIM is the most frequently used activity scale in the world in medical rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Gozde Iyigün, PhD, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, North Cyprus Via Mersin 10 Turkey, Cyprus